CLINICAL TRIAL: NCT03583489
Title: A Randomised, Double-blind, Placebo-controlled, Crossover Study in Healthy Adult Subjects to Investigate the Effect of Intravenous APD421, With and Without Ondansetron, on Cardiac Conduction
Brief Title: Study of APD421 With and Without Ondansetron
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acacia Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: DP10022
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- APD421 (Experimental)
  Interventions: Drug: APD421
- APD421 + ondansetron (Experimental)
  Interventions: Drug: APD421; Drug: Ondansetron

INTERVENTIONS:
Drug: APD421 — 10 mg IV
  Arms: APD421; APD421 + ondansetron
Drug: Placebo — IV
  Arms: Placebo
Drug: Ondansetron — 4 mg IV
  Arms: APD421 + ondansetron

SUMMARY:
Collection of pharmacokinetic and electrocardiograph data from healthy volunteers given APD421 +/- ondansetron

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects
2. Age 18 to 65 years of age at time of signing ICF
3. Body mass index (BMI) of 18 to 30 kg/m2
4. Must be willing and able to communicate and participate in the whole study
5. Must provide written informed consent
6. Must agree to use an adequate method of contraception

Exclusion Criteria:

1. Subjects who have received any investigational medicinal product (IMP) in a clinical research study within the 3 months prior to IMP administration on this study
2. Subjects who are study site employees, or immediate family members of a study site or sponsor employee
3. Subjects who have previously been enrolled in this study
4. Women who are pregnant or breastfeeding
5. Subjects who have received amisulpride for any indication within the previous 4 weeks
6. Allergy to amisulpride or any of the excipients of APD421 or ondansetron
7. History of any drug or alcohol abuse in the past 2 years
8. Regular alcohol consumption >21 units per week
9. Current smokers and those who have smoked within the last 12 months; this includes cigarettes, e-cigarettes and nicotine replacement products (current smoking may be assessed by a validated technique such as urine or serum cotinine levels)
10. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening
11. History of epilepsy
12. History of clinically significant syncope
13. Family history of sudden death
14. Family history of premature cardiovascular death
15. Clinically significant history or family history of congenital long QT syndrome (e.g. Romano-Ward syndrome, Jervell and Lange-Nielson syndrome) or Brugada's syndrome
16. History of clinically significant arrhythmias or ischaemic heart disease (especially ventricular arrhythmias, atrial fibrillation (AF), recent conversion from AF or coronary spasm)
17. Conditions predisposing the volunteer to electrolyte imbalances (e.g. altered nutritional states, chronic vomiting, anorexia nervosa, bulimia nervosa)
18. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG that may interfere with the interpretation of QTc interval changes.

    This includes subjects with any of the following at screening:
    * Absence of regular supraventricular rhythm
    * Clinically significant PR (PQ) interval prolongation
    * Intermittent second or third degree AV block
    * Incomplete or complete bundle branch block.
    * Abnormal T-wave morphology
    * Prolonged QTcB >450 ms or shortened QTcB < 350 ms or family history of long QT syndrome Subject with borderline deviations from these criteria may be included if the deviations do not pose a safety risk, as judged by the investigator
19. Clinically significant abnormal biochemistry, haematology or urinalysis at screening as judged by the investigator, especially:

    * Creatinine clearance (estimated using Cockcroft-Gault formula) < 60 mL/min
    * Alanine aminotransferase (ALT) > 1.5 x upper limit of normal or bilirubin > 3 x upper limit of normal
20. Positive drugs of abuse test result
21. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results at screening
22. Donation or loss of greater than 100 mL of blood within the 3 months prior to screening or planned blood donation during the study until after final visit
23. Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than 4 g per day paracetamol) or herbal remedies in the 14 days before IMP administration
24. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-13 (Actual)

PRIMARY OUTCOMES:
ddQTcF | 0-6 hours
  Placebo-corrected change-from-baseline QTcF interval

CONTACTS AND LOCATIONS:
Overall Officials: Muna Albayaty, Principal Investigator — Early Phase Clinical Unit
Locations (1):
- Early Phase Clinical Unit, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fox GM, Albayaty M, Walker JL, Xue H, Darpo B. Intravenous Amisulpride Does Not Meaningfully Prolong the QTc Interval at Doses Effective for the Management of Postoperative Nausea and Vomiting. Anesth Analg. 2021 Jan;132(1):150-159. doi: 10.1213/ANE.0000000000004538. PMID 31913911